CLINICAL TRIAL: NCT03750578
Title: Distraction in the Emergency Using Virtual Reality for Intravenous Needs in Children to Improve Comfort (DEVINCI): A Pilot Randomized Controlled Trial
Brief Title: Virtual Reality for Needle Procedures in the Pediatric Emergency Department
Acronym: DEVINCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Esli Osmanlliu, Fellow, Pediatric Emergency Medicine, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-2074
Record Dates: First submitted 2018-09-09; First posted 2018-11-23 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Procedural Anxiety; Pain
Keywords: virtual reality; procedural pain; pediatric emergency department; procedural anxiety
MeSH Terms: conditions — Pain; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Interventions. When venipuncture (either for IV line insertion or diagnostic venipuncture) is prescribed by a physician, a topical anesthetic cream (Maxilene® 4 - Lidocaine 4%) will be proposed to the patient, as standard of care. Usual positioning will be used by the staff nurse.
  A) Virtual reality: Patients in this group will be offered virtual reality distraction through the use of OR.
  B) Control intervention (standard of care): Patients in this group will receive standard care, including the proposition to use topical anesthetic cream prior to venipuncture attempt, usual distraction and positioning proposed by the treating nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Patients in this group will be offered virtual reality distraction through the use of OR in addition to standard of care.
  Interventions: Behavioral: Virtual Reality goggle (Oculus Rift ® Helmet)
- Standard of care group (No Intervention): Patients in this group will receive standard care, including the proposition to use topical anesthetic cream prior to venipuncture attempt, usual distraction and positioning proposed by the treating nurse.

INTERVENTIONS:
Behavioral: Virtual Reality goggle (Oculus Rift ® Helmet) — as described
  Arms: Virtual Reality Group

SUMMARY:
Venipuncture is a frequently performed painful and anxiogenic procedure in the paediatric emergency department (PED). Topical anesthetic creams are used to reduce pain, but additional modalities can modulate the nociceptive experience and distress associated with venipuncture. Distraction can improve a patient's experience by mitigating their ability to focus on the painful sensory input. Through its immersive nature, virtual reality (VR) has the potential to distract patients from a 'real world' negative experience such as venipuncture. Given the potential for short- and long-term consequences of poorly controlled pain and distress in children, healthcare professionals must optimize patient comfort during medically required procedures. The aim of this pilot pragmatic RCT study is to determine the feasibility, acceptability and preliminary effect of a VR device (head-mounted Oculus Rift® (OR)) for pain and distress reduction associated with venipuncture in the PED.

DETAILED DESCRIPTION:
INTRODUCTION Pain management of venipuncture in the Paediatric Emergency Department (PED)

Inadequate pain management in paediatrics is known to have significant short and long-term consequences, such as negative memories, and greater pain perception during future procedures. This can in turn lead to chronic healthcare avoidance, with potential implications for increased morbidity. Suboptimal comfort plan is still consistently reported in the literature Venipuncture is a frequently performed painful and anxiogenic procedure in the paediatric emergency department (PED). It is among the most important causes of pain in paediatric wards. This can be distressing for children, parents and healthcare workers (HCW). Indeed, venipuncture is the leading cause of pain among hospitalized children. Up to 51% of pre-adolescents reported high levels of distress associated with this procedure. Many children reported moderate to severe procedural pain during their hospitalization according to recent studies. Moreover, physiologic evidence of distress has been reported in caregivers as they witness ED-based venipuncture in their child. Improved pain and distress management during venipuncture can also significantly decrease distress in ED nurses performing the procedure. It is therefore imperative to minimize the pain and distress associated with venipuncture, especially in a stressful environment such as the PED. Therefore, multimodal approaches are proposed, with combined strategies such as the four essential components by Friedrichsdorf, which include the use of topical anaesthetics, sucrose in neonate, comfortable positioning and distraction.

Pharmacological intervention: Topical anesthetics To reduce the discomfort generated by a venipuncture, the use of a topical anaesthetic cream is recommended prior to needle procedures, with options including EMLA ®, amethocaine and lidocaine. These products have shown favourable results when the cream is applied prior to venipuncture and IV cannulation. In the department, this strategy was introduced in 2013 and is available through a collective order for nurses to use. The cream can be applied by a triage nurse suspecting that the child will require venipuncture, or by the physician whose management plan includes a needle puncture. Unfortunately, despite no real disadvantage to its application, this is a strategy often forgotten by the treating team. At the study institution, the investigators use Maxilene®. Its application is shorter than EMLA, only requiring a 30 minute wait, which is often less than the time lapse, in the study PED, between the prescription of a venipuncture and the actual intervention. Moreover, the anesthetic cream has been proven to improve procedure success on first attempt and to shorten procedure time, compared to placebo. Despite these advantages, this strategy remains scarcely used as mentioned above.

Physical intervention: Comfort Position Due to their developmental characteristics, it is often difficult for children to rationally understand the indication for venipuncture. Immobilization is therefore used in many instances - up to 74% of the time according to a previous report - for intravenous (IV) placement or blood procuration. However, child restrain should be avoided as much as possible. Despite the use of topical anesthetics, venipuncture remains a traumatic experience for many children who are restrained. For this reason, a sitting position is encouraged in the literature to increase the comfort of paediatric patients during venipuncture.

Psychological intervention: Distraction Given the significant distress associated with venipuncture despite improvement with the use of topical anesthetics and positioning, other psychological adjuncts to pain management are important components of pain and distress management related to needle procedures. Psychological interventions are recognized strategies for pain and distress management in this setting, given their simplicity, practicality, and at a relatively low cost. Side effects are usually absent to minimal. Distraction is one such modality, based on the gate control theory, which improves a patient's experience by mitigating their ability to focus on the painful sensory input. Modalities such as the hide and find games ''I spy'', video games, bubbles, cartoons, ''stress balls'', and other sensory modalities have been used as adjuncts to pain management during venipuncture in children. The choice of modality depends on the setting and on the child's developmental age. Effective distraction techniques focus on children empowerment through attention to their preferences, using either active (eg. electronic games, ''I spy'' games) or passive (eg. music, video on television or tablet) distraction. In the study department, distraction strategies have been improved in the recent years by the Equipe Analgésie Urgence (EAU) team creating giant hide and find games in the procedure rooms and introducing electronic tablets for use during procedures. Further, members of the study team also studied other interventions done to distract children during painful procedures.

Through its immersive nature, virtual reality (VR) has the potential to effectively distract patients from a ''real world'' negative experience such as venipuncture. It is hypothesized that VR produces analgesia through inter-cortical modulation, which may explain decreases in the pain matrix seen in functional magnetic resonance imaging of patients exposed to VR while experiencing painful procedures.

Virtual reality in the PED Immersive virtual reality has been documented in different settings, including burn units, hematology-oncology units, and orthopaedic procedural sedation. A recent randomized control trial (RCT) demonstrated a reduction of procedural pain and anxiety in patients 10-21 years old undergoing blood drawing at a phlebotomy outpatient clinic. In the care of burn patients, VR was shown to improve patient experience and clinical outcomes. To the investigators' knowledge there is no study on VR for procedural pain management in the PED.

A recent review of VR in paediatric patients describes it as "a promising new technology that offers unique opportunities to modulate the experience of pain''. Potential side effects are few and infrequent. These include visually induced motion sickness, a risk of collisions with the surrounding environment, and a potential for creating ''false memories'' in younger children. These potential side effects can be reduced by excluding younger children (<7 years old) until more suitable technologies are developed for this age group and also by working on the code source of a video (when possible) to modulate speed, pop ups, and other animations to better control for cyber-sicknesses.

Of note, the use of VR in healthcare settings has become more accessible due to the development of more portable and affordable systems. In this study, the investigators will use the Oculus Rift® (OR), which was purchased and mass produced by Facebook, allowing access to the latest technology in VR at a relatively low cost. OR is a VR tool that provides a wide field of view (FOV), high resolution display, integrated 3D audio and motion detection. In addition, its highly immersive properties could help achieve more distraction compared to other VR techniques as a review has shown that the sense of presence influences the effectiveness of VR-based analgesia. Presence refers to a subjective psychological state of consciousness of being in the virtual world. Immersiveness refers to the physical environment that could be quantified by measuring the field of view or the peripheral vision in the VR goggles.

The aims of this pilot RCT study is to address key areas (research design, methods, outcome measures, sample size, etc.) prior to conducting a future definitive trial. The investigators will therefore determine the acceptability and feasibility of a VR distraction using the OR in children requiring venipuncture in PED. The investigators also plan to evaluate the feasibility of the design and research methodology.

Objectives:

1. To determine the feasibility and acceptability of VR distraction using the OR in children undergoing venipuncture (IV line insertion or diagnostic venipuncture) in the PED.
2. To examine the preliminary effect of VR compared to standard practice on children's pain and distress related to venipuncture in the PED. Baseline estimate of the primary outcome (pain) will also inform sample size calculation of the definitive trial.
3. To determine parents', children's, and healthcare workers' (HCW) satisfaction regarding the use of VR for pain and distress management associated with venipuncture in the PED.
4. To determine feasibility and acceptability of the research design and methods including: recruitment rate, randomization and allocation, outcome measures, delivery of the interventions, rates of questionnaire completion, appropriateness of the inclusion criteria, among others.

METHODS. Design. Pilot pragmatic randomized control study using a parallel design with two groups: a) experimental group (VR+standard practice of needle-related pain management) or control (standard practice of needle-related pain management) Setting. The research will be conducted in a single ED, in a tertiary care paediatric university-affiliated hospital (Université de Montréal), the CHU Sainte-Justine in Montreal from August 2018 to June 2019. Sainte-Justine ED census is more than 80 000 patient-year.

Sample. Children from 7 to 17 years old who require venipuncture (IV line placement or diagnostic venipuncture) as prescribed by an attending physician. Research nurses and research assistants from the "Programme Intégré d'Étudiants à l'Urgence Volontaires pour la Recherche en Enfance de Sainte-Justine (PIEUVRES)" will identify eligible families in the waiting room of the ED using the institutional computerized database (between 8 AM and 8PM). These research assistants will approach a convenience sample of participants during day or evening shifts in the ED. Once they have accepted to participate and provided informed parent's consent and child's assent, participating families will be enrolled in the study.

As this is a pilot study, no sample size calculation is required. The investigators will randomize patients to one of the two intervention groups according to a list of randomization generated by an independent biostatistician. The investigators aim to recruit a total of 60 participants (30 patients/group) who will be randomized among the two groups during the study period. The investigators consider that this number would be adequate to provide information regarding feasibility of the intervention and study process/measures. It is estimated that close to 15 venipunctures are performed in the study department on a daily basis. The investigators therefore expect to reach the sample size within 9 months of the study start.

Interventions. When venipuncture (either for IV line insertion or diagnostic venipuncture) is prescribed by a physician, a topical anesthetic cream (Maxilene® 4 - Lidocaine 4%) will be proposed to the patient, as standard of care. Usual positioning will be used by the staff nurse.

A) RV : Patients in this group will be offered virtual reality distraction through the use of OR. VR produces a high level of immersion, with high photorealism while maintaining the low latency necessary to induce presence and prevent cyber-sickness symptoms such as nausea, vomiting, headache. The video game was developed by the study team with three levels of difficulty tailored to the children's developmental stages, and adapted to a hospital environment, allowing control over its components designed to maximize the feeling of immersion and minimize cyber-sickness symptoms. The game was approved by a team of healthcare professionals involved in paediatric care. The game, oculus goggles and computer will be available in the PED at the onset of the study. The oculus goggle will be adjusted to the head of each child randomized to this group before any procedure and a period of 3 minutes will be allotted prior to venipuncture. This will allow the child to get familiarized with the game and immersed in the virtual environment (See photos in Annex).

B) Control intervention (standard of care): Patients in this group will receive standard care, including the proposition to use topical anesthetic cream prior to venipuncture attempt, usual distraction and positioning proposed by the treating nurse. Standard behavioural techniques to relax children will be employed.

ELIGIBILITY:
Inclusion Criteria:

• Prescription of a venipuncture (IV line placement or diagnostic venipuncture) by an attending physician

Exclusion Criteria:

* Unstable patient or urgent procedure required
* Cognitive impairment that would render interaction with the VR game and/or answer to the study questionaires unfeasable.
* Diagnosis of epilepsy or any other condition precluding use of VR technology.
* A parent is unavailable to provide consent for participation in the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Self-reported pain during the procedure: Verbal Numerical Rating Scale (VNRS) | This outcome will be measured within 2 minutes of the end of the procedure (removal of needle/catheter from vein and of physical restraint in patients where it was used) by asking the child to rate their level of pain during the procedure.
  The primary outcome of this study is the mean pain score felt during the procedure (self-report of pain level during the procedure) measured by the Verbal Numerical Rating Scale (VNRS).
  The VNRS consists of pain scale from 0 (no pain) to 10 (extreme pain). It is a well-established, valid, and reliable tool for the self-report of pain intensity in children as young as 6 years of age. This scale is widely used as it requires a lower degree of abstraction and less resources when compared to the Visual Analog Scale (VAS). The VNRS requires no physical tools, which explains its wide use in older children and adults with acute pain.

SECONDARY OUTCOMES:
Evaluation of overall pain management during venipuncture, with respect to pain relief, side effects, physical recovery, and emotional recovery. | Measured within 5 minutes following the end procedure (removal of needle/catheter from vein and of physical restraint in patients where it was used)
  Individual 0 to 10 rating scales (without subscales), will be filled by the patient, parent and nurse present during the venipuncture.
  0 indicates "not at all", whereas 10 indicated "extremely" with respect to the question asked. Participants can only choose integers between 0 and 10.
  The results obtained from this scale aim to inform the study team on the participants' perception of pain management received by children undergoing a venipuncture, with respect to pain relief, side effects, physical recovery, and emotional recovery.
  The question asked is the following:
  "Considering pain relief, side effects, physical recovery, and emotional recovery, are you satisfied with the treatments your child received for pain? (0 = not at all, 10 = extremely)"
Hetero-evaluation (by research nurse) of procedure-related distress | Measured during the procedure (period between the start of physical restraint or needle/catheter insertion until needle/catheter removal from vein and end of physical restraint in patients where it was used)
  Will be measured with the Procedure Behaviour Check List (PBCL). Consists of 8 sub-categories, graded 1 (very light) to 5 (extremely intense), for maximum of 40 points. According to a systematic review of observational measures of pain in children and adolescents, this scale was among the scales with the best balance of evidence, ease of use, and validity for the evaluation for pain-related distress
Baseline pain score: Verbal Numerical Rating Scale (VNRS) | Measured following recruitment and at most 10 minutes before the start of the procedure (before the start of physical restraint or needle/catheter insertion)
  Self-report of pain level at baseline, measured by the Verbal Numerical Rating Scale (VNRS). 0 (no pain) to 10 (extreme pain) pain scale. The NRS is a well-established, valid, and reliable tool for the self-report of pain intensity in children as young as 6 years of age. This scale is widely used as it requires a lower degree of abstraction and less resources when compared to the VAS. The VNRS is even simpler, as it requires no physical tools, which explains its wide use in older children and adults with acute pain.
Auto-evaluation of post procedure-related distress | Measured within 5 minutes following the end of the procedure (removal of needle/catheter from vein and of physical restraint in patients where it was used)
  Measured with the Child Fear Scale (CFS), a self-reported measure of anxiety adapted from the Faces Anxiety Scale (McKinley et al., 2003) for specific use in children undergoing painful experiences. It presents five faces ranging from 0 (no fear) through 4 (extremely fearful). The child is asked to indicate which face shows best how he/she feels during the procedure.
Auto-evaluation of baseline procedure-related distress | Measured following recruitment and at most 10 minutes before the start of the procedure (before the start of physical restraint or needle/catheter insertion)
  Measured with the Child Fear Scale (CFS), a self-reported measure of anxiety adapted from the Faces Anxiety Scale (McKinley et al., 2003) for specific use in children undergoing painful experiences. It presents five faces ranging from 0 (no fear) through 4 (extremely fearful). The child is asked to indicate which face shows best how he/she feels during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Esli Osmanlliu, MD,FRCPC, Principal Investigator — Emergency Department, UdM; Evelyne D. Trottier, MD,FRCPC, Study Director — Emergency Department, UdM; Sylvie Lemay, PhD, Study Director — CHU Sainte-Justine Research Centre
Locations (1):
- St Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali S, Chambers A, Johnson DW, Newton AS, Vandermeer B, Williamson J, Curtis SJ. Reported practice variation in pediatric pain management: a survey of Canadian pediatric emergency physicians. CJEM. 2014 Sep;16(5):352-60. doi: 10.2310/8000.2013.131261. PMID 25227643
- [Background] Ali S, McGrath T, Drendel AL. An Evidence-Based Approach to Minimizing Acute Procedural Pain in the Emergency Department and Beyond. Pediatr Emerg Care. 2016 Jan;32(1):36-42; quiz 43-4. doi: 10.1097/PEC.0000000000000669. PMID 26720064
- [Background] American Academy of Pediatrics; Committee on Fetus and Newborn; Canadian Paediatric Society; Fetus and Newborn Committee. Prevention and management of pain in the neonate. An update. Adv Neonatal Care. 2007 Jun;7(3):151-60. doi: 10.1097/01.anc.0000278214.49133.7d. PMID 17844779
- [Background] American Academy of Pediatrics. Committee on Psychosocial Aspects of Child and Family Health; Task Force on Pain in Infants, Children, and Adolescents. The assessment and management of acute pain in infants, children, and adolescents. Pediatrics. 2001 Sep;108(3):793-7. doi: 10.1542/peds.108.3.793. PMID 11533354
- [Background] Bailey B, Bergeron S, Gravel J, Daoust R. Comparison of four pain scales in children with acute abdominal pain in a pediatric emergency department. Ann Emerg Med. 2007 Oct;50(4):379-83, 383.e1-2. doi: 10.1016/j.annemergmed.2007.04.021. Epub 2007 Jun 22. PMID 17588706
- [Background] Bailey B, Daoust R, Doyon-Trottier E, Dauphin-Pierre S, Gravel J. Validation and properties of the verbal numeric scale in children with acute pain. Pain. 2010 May;149(2):216-221. doi: 10.1016/j.pain.2009.12.008. Epub 2010 Feb 25. PMID 20188471
- [Background] Bray L, Snodin J, Carter B. Holding and restraining children for clinical procedures within an acute care setting: an ethical consideration of the evidence. Nurs Inq. 2015 Jun;22(2):157-67. doi: 10.1111/nin.12074. Epub 2014 Jul 23. PMID 25053126
- [Background] Castarlenas E, Jensen MP, von Baeyer CL, Miro J. Psychometric Properties of the Numerical Rating Scale to Assess Self-Reported Pain Intensity in Children and Adolescents: A Systematic Review. Clin J Pain. 2017 Apr;33(4):376-383. doi: 10.1097/AJP.0000000000000406. PMID 27518484
- [Background] Chen E, Zeltzer LK, Craske MG, Katz ER. Children's memories for painful cancer treatment procedures: implications for distress. Child Dev. 2000 Jul-Aug;71(4):933-47. doi: 10.1111/1467-8624.00200. PMID 11016557
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Fein JA, Zempsky WT, Cravero JP; Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine; American Academy of Pediatrics. Relief of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 2012 Nov;130(5):e1391-405. doi: 10.1542/peds.2012-2536. Epub 2012 Oct 29. PMID 23109683
- [Background] Foster JP, Taylor C, Spence K. Topical anaesthesia for needle-related pain in newborn infants. Cochrane Database Syst Rev. 2017 Feb 4;2(2):CD010331. doi: 10.1002/14651858.CD010331.pub2. PMID 28160271
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Humphrey GB, Boon CM, van Linden van den Heuvell GF, van de Wiel HB. The occurrence of high levels of acute behavioral distress in children and adolescents undergoing routine venipunctures. Pediatrics. 1992 Jul;90(1 Pt 1):87-91. PMID 1614786
- [Background] Kennedy RM, Luhmann J, Zempsky WT. Clinical implications of unmanaged needle-insertion pain and distress in children. Pediatrics. 2008 Nov;122 Suppl 3:S130-3. doi: 10.1542/peds.2008-1055e. PMID 18978006
- [Background] Lacey CM, Finkelstein M, Thygeson MV. The impact of positioning on fear during immunizations: supine versus sitting up. J Pediatr Nurs. 2008 Jun;23(3):195-200. doi: 10.1016/j.pedn.2007.09.007. PMID 18492548
- [Background] LeBaron S, Zeltzer L. Assessment of acute pain and anxiety in children and adolescents by self-reports, observer reports, and a behavior checklist. J Consult Clin Psychol. 1984 Oct;52(5):729-38. doi: 10.1037//0022-006x.52.5.729. No abstract available. PMID 6501658
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Rogers TL, Ostrow CL. The use of EMLA cream to decrease venipuncture pain in children. J Pediatr Nurs. 2004 Feb;19(1):33-9. doi: 10.1016/j.pedn.2003.09.005. PMID 14963868
- [Background] Sanchez-Rodriguez E, Miro J, Castarlenas E. A comparison of four self-report scales of pain intensity in 6- to 8-year-old children. Pain. 2012 Aug;153(8):1715-1719. doi: 10.1016/j.pain.2012.05.007. Epub 2012 Jun 15. PMID 22703691
- [Background] Svendsen EJ, Pedersen R, Moen A, Bjork IT. Exploring perspectives on restraint during medical procedures in paediatric care: a qualitative interview study with nurses and physicians. Int J Qual Stud Health Well-being. 2017 Dec;12(1):1363623. doi: 10.1080/17482631.2017.1363623. PMID 28889788
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline (summary). CMAJ. 2010 Dec 14;182(18):1989-95. doi: 10.1503/cmaj.092048. Epub 2010 Nov 22. No abstract available. PMID 21098067
- [Background] Taylor EM, Boyer K, Campbell FA. Pain in hospitalized children: a prospective cross-sectional survey of pain prevalence, intensity, assessment and management in a Canadian pediatric teaching hospital. Pain Res Manag. 2008 Jan-Feb;13(1):25-32. doi: 10.1155/2008/478102. PMID 18301813
- [Background] Tsze DS, von Baeyer CL, Pahalyants V, Dayan PS. Validity and Reliability of the Verbal Numerical Rating Scale for Children Aged 4 to 17 Years With Acute Pain. Ann Emerg Med. 2018 Jun;71(6):691-702.e3. doi: 10.1016/j.annemergmed.2017.09.009. Epub 2017 Nov 6. PMID 29107409
- [Background] Van Hulle Vincent C. Nurses' perceptions of children's pain: a pilot study of cognitive representations. J Pain Symptom Manage. 2007 Mar;33(3):290-301. doi: 10.1016/j.jpainsymman.2006.08.008. PMID 17349498
- [Background] Weisman SJ, Bernstein B, Schechter NL. Consequences of inadequate analgesia during painful procedures in children. Arch Pediatr Adolesc Med. 1998 Feb;152(2):147-9. doi: 10.1001/archpedi.152.2.147. PMID 9491040
- [Background] Wente SJ. Nonpharmacologic pediatric pain management in emergency departments: a systematic review of the literature. J Emerg Nurs. 2013 Mar;39(2):140-50. doi: 10.1016/j.jen.2012.09.011. Epub 2012 Nov 28. PMID 23199786
- [Derived] Osmanlliu E, Trottier ED, Bailey B, Lagace M, Certain M, Khadra C, Sanchez M, Theriault C, Paquin D, Cotes-Turpin C, Le May S. Distraction in the Emergency department using Virtual reality for INtravenous procedures in Children to Improve comfort (DEVINCI): a pilot pragmatic randomized controlled trial. CJEM. 2021 Jan;23(1):94-102. doi: 10.1007/s43678-020-00006-6. Epub 2020 Dec 23. PMID 33683617